CLINICAL TRIAL: NCT07367165
Title: Improving Palatal Donor Site Healing and Reducing Postoperative Morbidity With Concentrated Growth Factor and Collagen Fleece: Randomized Controlled Clinical Study
Brief Title: Effects of CGF and Collagen Fleece on Palatal Donor Site Healing: A Randomized Clinical Trial
Acronym: PAL-HEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Cuneyt Asim Aral, Professor of Periodontology, Inonu University Faculty of Dentistry, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUCREC.2023.82; TDH-2024-3515 (Other Grant/Funding Number: Inönü University Scientific Research Projects Coordination Office)
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Wound Healing
Keywords: Concentrated Growth Factor (CGF); Collagen Fleece; Palatal Donor Site; Soft Tissue Graft Harvesting; Wound Healing; Oral Soft Tissue Regeneration; Postoperative Morbidity; Gingival Thickness; Periodontal Plastic Surgery; Autogenous Graft
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of three parallel intervention arms:
  1. a Concentrated Growth Factor (CGF) group,
  2. a Collagen Fleece (CF) group, and
  3. a control group receiving a collagen sponge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concentrated Growth Factor (CGF) (Experimental)
  Interventions: Biological: Concentrated Growth Factor (CGF)
- Collagen Fleece (CF) (Experimental)
  Interventions: Biological: Collagen Fleece (CF)
- Control (Collagen Sponge) (Experimental)
  Interventions: Biological: Collagen Sponge (Control)

INTERVENTIONS:
Biological: Concentrated Growth Factor (CGF) — A CGF membrane prepared from the participant's venous blood was applied to the palatal donor site following soft tissue graft harvesting. The membrane was stabilized using sutures and covered with an oral wound dressing to support healing and reduce postoperative morbidity.
  Arms: Concentrated Growth Factor (CGF)
Biological: Collagen Fleece (CF) — A collagen fleece was placed over the palatal donor site immediately after tissue harvesting. The material was stabilized with sutures and covered with an oral wound dressing to promote donor site healing.
  Arms: Collagen Fleece (CF)
Biological: Collagen Sponge (Control) — A sterile collagen sponge was applied to the palatal donor site as the control intervention. The sponge was secured with sutures and covered with an oral wound dressing, serving as the standard healing approach.
  Arms: Control (Collagen Sponge)

SUMMARY:
This study investigated whether applying Concentrated Growth Factor (CGF) or Collagen Fleece (CF) to the palatal donor site after autogenous soft tissue graft harvesting could improve wound healing and reduce postoperative discomfort. The palatal donor site often requires several weeks to heal, and patients may experience pain, delayed epithelialization, and difficulty in daily oral functions. Biologically active materials such as CGF and collagen-based dressings may help accelerate tissue repair and improve patient comfort.

A total of 38 systemically healthy adults requiring soft tissue graft harvesting were enrolled and assigned to three groups: CGF, CF, or control. In all groups, the applied material was stabilized with sutures and covered with an oral wound dressing. Palatal tissue thickness was measured at baseline and at 1, 3, and 6 months. Wound healing was evaluated on postoperative days 3, 7, and 14 and at 1 month using standardized clinical indices. Patient-reported outcomes, including pain, analgesic use, and oral health-related quality of life, were also recorded.

The study aims to determine whether CGF or CF provides superior healing, better preservation of palatal tissue thickness, and reduced postoperative morbidity compared with spontaneous healing. Findings from this trial may help clinicians select supportive materials that enhance donor-site healing and improve patient comfort after periodontal soft tissue graft procedures.

DETAILED DESCRIPTION:
Autogenous soft tissue grafts harvested from the palatal mucosa remain the gold standard for increasing keratinized tissue width and augmenting gingival thickness in periodontal and peri-implant plastic surgery. Despite their predictable clinical benefits, palatal donor sites frequently exhibit delayed epithelialization, postoperative bleeding, pain, and functional discomfort. These factors contribute to increased morbidity and may negatively affect patient compliance and overall satisfaction with periodontal treatment.

Recent biomaterials such as Concentrated Growth Factor (CGF) and collagen-based dressings have been proposed to enhance soft tissue regeneration and accelerate wound healing. CGF is produced by centrifugation of autologous blood and contains a dense fibrin matrix enriched with platelets, leukocytes, and growth factors. Its biological profile has been associated with improved angiogenesis, fibroblast migration, and soft-tissue remodeling. Collagen fleece (CF), a widely used resorbable matrix, provides hemostasis, a physical barrier for wound protection, and a scaffold that supports early epithelial migration. However, the comparative clinical efficacy of CGF and CF on palatal donor site healing has not been clearly established in controlled human studies.

This randomized controlled clinical trial was designed to evaluate the effects of CGF and CF on wound healing dynamics, preservation of palatal tissue thickness, and postoperative morbidity following standardized soft tissue graft harvesting. Thirty-eight systemically healthy adult patients requiring autogenous grafts were included and allocated to one of three groups: CGF, CF, or control. In the test groups, either CGF or CF was applied to the donor site, stabilized with sutures, and covered with an oral wound dressing. In the control group, a collagen sponge was placed beneath the wound dressing. All groups received identical postoperative care.

Primary and secondary outcome measures included changes in palatal tissue thickness, wound healing scores, epithelialization patterns, patient-reported pain levels, analgesic consumption, bleeding, and oral health-related quality of life. Tissue thickness was evaluated at baseline and at 1, 3, and 6 months postoperatively. Wound healing characteristics were recorded on postoperative days 3, 7, and 14, and at 1 month, using standardized indices such as the H₂O₂ bubbling test, the Modified Manchester Scar Scale, and the Landry-Turnbull-Howley healing index. Pain intensity and functional discomfort were assessed using visual analog scales (VAS), while overall patient impact was measured with the OHIP-14 questionnaire.

The central hypothesis of this study was that both CGF and CF would enhance palatal donor site healing relative to spontaneous healing, and that CGF would demonstrate additional benefits due to its autologous biological activity. The findings of this trial are expected to provide clinicians with evidence-based guidance on the use of supportive biomaterials to reduce postoperative morbidity, improve patient comfort, and optimize regenerative outcomes after periodontal soft-tissue grafting procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Systemically healthy individuals
* Good oral hygiene
* Stable periodontal condition
* Indication for mucogingival surgery requiring autogenous soft tissue grafting
* Free gingival graft or de-epithelialized free gingival graft combined with either a coronally advanced flap or tunnel technique

Exclusion Criteria:

* Smoking
* Pregnancy or lactation
* Systemic diseases affecting wound healing
* Use of medications known to interfere with healing
* History of radiotherapy or chemotherapy
* Poor oral hygiene or uncontrolled periodontal disease
* Concomitant bone surgery or implant placement
* Surgical duration exceeding 2 hours

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Change in Palatal Tissue Thickness at the Donor Site | Baseline, 1 month, 3 months, and 6 months postoperatively
  Palatal tissue thickness at the donor site was measured using a standardized periodontal probe and/or caliper at baseline and during follow-up. Changes in thickness were compared among the CGF, CF, and control groups to assess the effectiveness of each intervention in maintaining palatal tissue thickness.

SECONDARY OUTCOMES:
Re-epithelialization Assessed by H₂O₂ Bubbling Test | Postoperative Day 3, Day 7, Day 14, and 1 Month
  Re-epithelialization of the palatal donor site was evaluated using the hydrogen peroxide (H₂O₂) bubbling test. The presence or absence of bubbling indicated incomplete or complete epithelial coverage. Healing progression was compared among the three groups.
Wound Healing Quality - Landry-Turnbull-Howley (LTH) Index | Postoperative Day 7, Day 14, and 1 Month
  Wound healing at the palatal donor site was assessed using the Landry-Turnbull-Howley (LTH) Wound Healing Index, a clinician-rated ordinal scale evaluating overall soft tissue healing based on tissue color, bleeding on palpation, presence of granulation tissue, epithelialization of the incision margin, and suppuration.
  Healing is scored on a 5-point scale ranging from 1 to 5, where:
  1. = very poor,
  2. = poor,
  3. = good,
  4. = very good,
  5. = excellent.
  The total score therefore ranges from 1 (worst healing) to 5 (best healing), with higher scores indicating better wound healing and more favorable clinical outcomes.
Scar Formation - Modified Manchester Scar Scale (MSS) | Postoperative Day 7, Day 14, and 1 Month
  Scar appearance at the palatal donor site was evaluated using the Modified Manchester Scar Scale (MSS), a clinician-rated scale assessing color, contour, and distortion. Each parameter is scored from 0 to 2 (0 = normal/best appearance, 2 = marked discrepancy/worst appearance), resulting in a total score range of 0-6. Lower scores indicate better scar quality and more favorable healing, whereas higher scores indicate poorer scar appearance. Assessments were performed at 1 and 3 months postoperatively.
Postoperative Pain - Visual Analog Scale (VAS) | Postoperative Day 1, Day 3, Day 7, Day 14
  Postoperative pain intensity was assessed using the Visual Analog Scale (VAS), a validated self-reported measure of subjective pain. Patients rated their pain on a 10-point scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores therefore represent greater pain severity and worse clinical outcomes. Pain scores were recorded at predefined postoperative intervals to monitor changes in pain intensity over time.
Analgesic Consumption | First 7 Days Postoperatively
  The total number of analgesic tablets consumed by each participant during the postoperative period was recorded to assess the need for pain control. Lower consumption indicates reduced postoperative morbidity.
Patient-Reported Oral Health-Related Quality of Life (OHIP-14) | Assessments were performed on postoperative days 3, 7 and 14.
  Oral health-related quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14), a validated patient-reported questionnaire consisting of 14 items across seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap.
  Each item is scored on a 5-point Likert scale (0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, 4 = very often). The total score ranges from 0 to 56, with higher scores indicating worse oral health-related quality of life and greater functional impairment, whereas lower scores reflect better patient-reported outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Inönü University Faculty of Dentistry, Department of Periodontology, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zucchelli G, Mounssif I. Periodontal plastic surgery. Periodontol 2000. 2015 Jun;68(1):333-68. doi: 10.1111/prd.12059. PMID 25867992
- [Background] Tavelli L, Barootchi S, Stefanini M, Zucchelli G, Giannobile WV, Wang HL. Wound healing dynamics, morbidity, and complications of palatal soft-tissue harvesting. Periodontol 2000. 2023 Jun;92(1):90-119. doi: 10.1111/prd.12466. Epub 2022 Dec 30. PMID 36583690
- [Background] Oliveira JA, da Silveira MI, Soares LFF, Alves RO, Carrera TMI, Azevedo MR, Oliveira GJPL, Pigossi SC. Wound-healing agents for palatal donor area: A network meta-analysis. Clin Oral Implants Res. 2024 Apr;35(4):359-376. doi: 10.1111/clr.14241. Epub 2024 Feb 5. PMID 38315151
- [Background] Lacoste E, Martineau I, Gagnon G. Platelet concentrates: effects of calcium and thrombin on endothelial cell proliferation and growth factor release. J Periodontol. 2003 Oct;74(10):1498-507. doi: 10.1902/jop.2003.74.10.1498. PMID 14653397
- [Background] Masuki H, Okudera T, Watanebe T, Suzuki M, Nishiyama K, Okudera H, Nakata K, Uematsu K, Su CY, Kawase T. Growth factor and pro-inflammatory cytokine contents in platelet-rich plasma (PRP), plasma rich in growth factors (PRGF), advanced platelet-rich fibrin (A-PRF), and concentrated growth factors (CGF). Int J Implant Dent. 2016 Dec;2(1):19. doi: 10.1186/s40729-016-0052-4. Epub 2016 Aug 22. PMID 27747711
- [Background] Li G, Wang H. Novel Applications of Concentrated Growth Factors in Facial Rejuvenation and Plastic Surgery. Facial Plast Surg. 2024 Feb;40(1):112-119. doi: 10.1055/a-1987-3459. Epub 2022 Nov 24. PMID 36423628
- [Background] Voormolen JH, Ringers J, Bots GT, van der Heide A, Hermans J. Hemostatic agents: brain tissue reaction and effectiveness. A comparative animal study using collagen fleece and oxidized cellulose. Neurosurgery. 1987 May;20(5):702-9. doi: 10.1227/00006123-198705000-00005. PMID 3601016
- [Background] Bienz SP, Gadzo N, Zuercher AN, Wiedemeier D, Jung RE, Thoma DS. Clinical and histological wound healing patterns of collagen-based substitutes: An experimental randomized controlled trial in standardized palatal defects in humans. J Clin Periodontol. 2024 Mar;51(3):319-329. doi: 10.1111/jcpe.13903. Epub 2023 Nov 28. PMID 38017650
- [Background] Zhang T, Yuan M, Hao X, Gao H, Teng M, Hu F, Liang Y, Deng J, Li F. Innovative biomaterials in promoting intraoral wound healing: Mechanisms, applications, and challenges. Mater Today Bio. 2025 Oct 28;35:102470. doi: 10.1016/j.mtbio.2025.102470. eCollection 2025 Dec. PMID 41255422
- [Background] Basma HS, Saleh MHA, Abou-Arraj RV, Imbrogno M, Ravida A, Wang HL, Li P, Geurs N. Patient-reported outcomes of palatal donor site healing using four different wound dressing modalities following free epithelialized mucosal grafts: A four-arm randomized controlled clinical trial. J Periodontol. 2023 Jan;94(1):88-97. doi: 10.1002/JPER.22-0172. Epub 2022 Aug 3. PMID 35754198